CLINICAL TRIAL: NCT04625127
Title: GaitBetter: Motor and Cognitive Training for Gait Rehabilitation and Falls Prevention in Stroke Survivors.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: GoldenGait LTD (Unknown)
Responsible Party: Principal Investigator, Paolo Bonato, Principal Investigator, Director of the Motion Analysis Laboratory, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020P002544
Record Dates: First submitted 2020-10-27; First posted 2020-11-12 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Stroke; Gait, Hemiplegic; Hemiplegia
Keywords: Stroke; Gait; Falls
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic; Hemiplegia | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Aim 2: Efficacy of the GaitBetter to improve motor-cognitive function of chronic stroke survivors (Experimental): The investigators propose a single-arm, non-randomized study to test the hypothesis that the GaitBetter training is effective in improving gait and cognition in individuals with chronic stroke. This design was chosen given the expected stability of functional recovery in this population.
  Interventions: Device: Treadmill gait training with GaitBetter
- Aim 3: Efficacy of the GaitBetter to improve rehabilitation outcomes in sub-acute stroke survivors (Experimental): The investigators propose a randomized, controlled study to evaluate the effects of using the GaitBetter system in patients with subacute stroke on recovery trajectory.
  Interventions: Other: Treadmill gait training with GaitBetter + Standard of care; Other: Standard of care

INTERVENTIONS:
Device: Treadmill gait training with GaitBetter — Participants will receive gait training with the GaitBetter solution for a total of 15 sessions (3 days a week for 5 weeks) each lasting approximately 45 minutes.
  Arms: Aim 2: Efficacy of the GaitBetter to improve motor-cognitive function of chronic stroke survivors
Other: Treadmill gait training with GaitBetter + Standard of care — Participants will receive gait training with the GaitBetter solution for a total of 15 sessions (3 days a week for 5 weeks) each lasting approximately 45 minutes. In addition, the investigators will record the number and duration of therapy sessions followed by the participant during standard of care.
  Arms: Aim 3: Efficacy of the GaitBetter to improve rehabilitation outcomes in sub-acute stroke survivors
Other: Standard of care — Participants will follow their standard of care. The investigators will record the number and duration of therapy sessions followed during standard of care.
  Arms: Aim 3: Efficacy of the GaitBetter to improve rehabilitation outcomes in sub-acute stroke survivors

SUMMARY:
In this research study, the investigators aim to test the usability and efficacy of the GaitBetter system for gait rehabilitation after stroke.

DETAILED DESCRIPTION:
This study consists of 3 distinct aims:

In Aim 1, the investigators will evaluate clinical acceptance of the GaitBetter solution by subjects and therapists. To do so, the investigators will run a pilot study to gather feedback from stakeholders (not reported here).

In Aim 2, the investigators will evaluate the efficacy of using the GaitBetter solution to improve motor-cognitive function of chronic stroke survivors. To do so, the investigators will run a single-arm, non-randomized study to test the hypothesis that the GaitBetter training is effective in improving gait and cognition in individuals with chronic stroke.

In Aim 3, the investigators will explore the efficacy of using the GaitBetter solution for improving rehabilitation outcomes in sub-acute stroke survivors. To do so, the investigators will run a randomized, controlled study to evaluate the effects of using the GaitBetter system in patients with subacute stroke on recovery trajectory.

ELIGIBILITY:
Inclusion Criteria:

* Male and females of age between 18 to 85 year of age
* History of one-sided ischemic or hemorrhagic stroke

  * Chronic: more than 6 months post-stroke (Aim 1 and Aim 2)
  * Subacute: within 8 weeks post-stroke (Aim 1 and Aim 3)
* Residual functional impairment of a lower extremity as a result of the stroke
* Ability to walk at least 15 meters with or without assistive devices (FIM walk subsection, levels 6 and 7)
* Ability to walk 3 consecutive minutes (5 minutes for Aim 2) on a treadmill at a speed equal to or greater than 0.22 m/s (0.8 km/h or 0.5 mph) with or without hand support.
* Medical clearance received from treating physician to participate in the gait training program proposed in the study

Exclusion Criteria:

* Severe aphasia limiting the ability to express needs or discomfort verbally or non-verbally
* Cognitive impairment limiting the ability to understand and follow instructions (as assessed by a score <23 on the Mini Mental State Examination)
* Previous diagnosis of neurological diseases other than stroke
* Recent history of lower extremity fractures (<12 months ago), unhealed wounds
* Current indication for isolation precautions (e.g. MRSA, VRE, C. difficile, and others)
* Severe visual impairments (as assessed by the NIH Stroke Scale Visual Field subscale. score >0)
* Hemispatial neglect (as assessed by the Line Bisection Test)
* Subjects diagnosed with a medical condition that would interfere with their participation in regular sustained exercise (such as a severe pulmonary and/or cardiovascular condition)
* For Aim 2: currently participating in a gait training intervention (PT or research)
* Adults with impaired decision-making capacity
* Women who are pregnant

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2021-07-23 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
10 meter walk test (in chronic stroke survivors, Aim 2) | Change from baseline scores at post-intervention (after 5 weeks)
  Evaluation of gait speed of chronic stroke survivors, in meters per second
10 meter walk test (in subacute stroke survivors, Aim 3) | Change from baseline scores at post-intervention (after 5 weeks)
  Evaluation of gait speed of subacute stroke survivors, in meters per second
Trail making test (in chronic stroke survivors, Aim 2) | Change from baseline scores at post-intervention (after 5 weeks)
  Evaluation of cognition status, in chronic stroke survivors. The test record the time to accomplish the task (higher values indicate slower performance)
Trail making test (in subacute stroke survivors, Aim 3) | Change from baseline scores at post-intervention (after 5 weeks)
  Evaluation of cognition status, in subacute stroke survivors. The test record the time to accomplish the task (higher values indicate slower performance)
Balance Evaluation Systems Test (mini-BESTest, in chronic stroke survivors, Aim 2) | Change from baseline scores at post-intervention (after 5 weeks)
  Comprehensive evaluation of balance and falls risks in chronic stroke survivors. Score from 0 to 108. Higher scores are reflecting better balance
Aim 3: Balance Evaluation Systems Test (mini-BESTest, in subacute stroke survivors, Aim 3) | Change from baseline scores at post-intervention (after 5 weeks)
  Comprehensive evaluation of balance and falls risks in subacute stroke survivors. Score from 0 to108. Higher scores are reflecting better balance

SECONDARY OUTCOMES:
Step length (in chronic stroke survivors, Aim 2) | Change from baseline scores at post-intervention (after 5 weeks)
  Evaluation of gait step length in chronic stroke survivors with an 3D motion capture system (in meters)
Step length (in subacute stroke survivors, Aim 3) | Change from baseline scores at post-intervention (after 5 weeks)
  Evaluation of gait step length in subacute stroke survivors with an 3D motion capture system (in meters)
Step width (in chronic stroke survivors, Aim 2) | Change from baseline scores at post-intervention (after 5 weeks)
  Evaluation of gait step width in chronic stroke survivors with an 3D motion capture system (in meters)
Step width (in subacute stroke survivors, Aim 3) | Change from baseline scores at post-intervention (after 5 weeks)
  Evaluation of gait step width in subacute stroke survivors with an 3D motion capture system (in meters)
Step symmetry (in chronic stroke survivors, Aim 2) | Change from baseline scores at post-intervention (after 5 weeks)
  Evaluation of gait step symmetry in chronic stroke survivors with an 3D motion capture system (ratio between paretic and non-paretic leg)
Step symmetry (in subacute stroke survivors, Aim 3) | Change from baseline scores at post-intervention (after 5 weeks)
  Evaluation of gait step symmetry in subacute stroke survivors with an 3D motion capture system (ratio between paretic and non-paretic leg)
Stance time (in chronic stroke survivors, Aim 2) | Change from baseline scores at post-intervention (after 5 weeks)
  Evaluation of gait stance time in chronic stroke survivors with an 3D motion capture system (in seconds)
Stance time (in subacute stroke survivors, Aim 3) | Change from baseline scores at post-intervention (after 5 weeks)
  Evaluation of gait stance time in subacute stroke survivors with an 3D motion capture system (in seconds)
Swing time (in chronic stroke survivors, Aim 2) | Change from baseline scores at post-intervention (after 5 weeks)
  Evaluation of gait swing time in chronic stroke survivors with an 3D motion capture system (in seconds)
Swing time (in subacute stroke survivors, Aim 3) | Change from baseline scores at post-intervention (after 5 weeks)
  Evaluation of gait swing time in subacute stroke survivors with an 3D motion capture system (in seconds)

OTHER OUTCOMES:
Montreal Cognitive Assessment (MoCA) (in chronic stroke survivors, Aim 2) | Change from baseline scores at post-intervention (after 5 weeks)
  Measure of the cognitive status in chronic stroke survivors
Montreal Cognitive Assessment (MoCA) (in subacute stroke survivors, Aim 3) | Change from baseline scores at post-intervention (after 5 weeks)
  Measure of the cognitive status in subacute stroke survivors
Symbol-Digit Modalities Test (SDMT) (in subacute stroke survivors, Aim 2) | Change from baseline scores at post-intervention (after 5 weeks)
  Measure of the cognitive status in chronic stroke survivors
Symbol-Digit Modalities Test (SDMT) (in subacute stroke survivors, Aim 3) | Change from baseline scores at post-intervention (after 5 weeks)
  Measure of the cognitive status in subacute stroke survivors
Hopkins Verbal Learning Test (Revised) (in chronic stroke survivors, Aim 2) | Change from baseline scores at post-intervention (after 5 weeks)
  Measure of the cognitive status in chronic stroke survivors
Hopkins Verbal Learning Test (Revised) (in subacute stroke survivors, Aim 3) | Change from baseline scores at post-intervention (after 5 weeks)
  Measure of the cognitive status in subacute stroke survivors
2-minutes walk test (2mwt) (in chronic stroke survivors, Aim 2) | Change from baseline scores at post-intervention (after 5 weeks)
  Measure of the gait endurance in chronic stroke survivors
2-minutes walk test (2mwt) (in subacute stroke survivors, Aim 3) | Change from baseline scores at post-intervention (after 5 weeks)
  Measure of the gait endurance in subacute stroke survivors
Functional Gait Assessment (FGA) (in chronic stroke survivors, Aim 2) | Change from baseline scores at post-intervention (after 5 weeks)
  Measure of the gait mobility, balance and falls risks in chronic stroke survivors
Functional Gait Assessment (FGA) (in subacute stroke survivors, Aim 3) | Change from baseline scores at post-intervention (after 5 weeks)
  Measure of the gait mobility, balance and falls risks in subacute stroke survivors
12-Item Short Form Health Survey (SF-12) (in chronic stroke survivors, Aim 2) | Change from baseline scores at post-intervention (after 5 weeks)
  Self-reported measure of quality of life
12-Item Short Form Health Survey (SF-12) (in subacute stroke survivors, Aim 3) | Change from baseline scores at post-intervention (after 5 weeks)
  Self-reported measure of quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bonato, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (1):
- Spaulding Rehabilitation Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No